CLINICAL TRIAL: NCT01021384
Title: Supporting the Well Being of Families of Young Children With Autism Spectrum
Brief Title: Supporting the Well Being of Families of Young Children With Autism Spectrum Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily Feinberg, Associate Professor, Boston Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-28799
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Maternal Depression
Keywords: Depression,; Early Intervention,; Behavior Disorder,; Parenting Skills,; Children with Special Health Care Needs,; Developmental Disabilities,; Family Support Programs
MeSH Terms: conditions — Depression; Mental Disorders; Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Problem Solving Education (Other)
  Interventions: Behavioral: Problem Solving Education

INTERVENTIONS:
Behavioral: Problem Solving Education — Problem Solving Education (PSE) is an evidenced-based empowerment strategy, targeted to mothers of young children to promote family well-being by decreasing the burden of maternal depressive symptoms and maternal parenting stress and improving social functioning.

SUMMARY:
The objective of this 2 year research project is to determine whether an evidenced-based empowerment strategy, Problem Solving Education (PSE), targeted to mothers of young children with autism spectrum disorders (ASDs), promotes family well-being by decreasing the burden of maternal depressive symptoms and maternal parenting stress and improving social functioning. We propose a randomized control trial involving 140 mothers who have children <4 years with confirmed ASDs. Based on the paradigm of the IOM report on mental health prevention research that highlights the importance of targeting interventions to at-risk populations who may not meet diagnostic criteria, all mothers of young children with ASDs will be eligible to participate. Consistent with previous studies of cognitive-behavioral interventions, the mother-child pairs will be followed for 9 months. The intervention will be embedded in two settings that provide services to young children with ASDs - Early Intervention (EI) programs and specialty developmental assessment clinics. We aim to support families during a critical juncture - when they are confronted with a new diagnosis and are asked to navigate a complex service system on their children's behalf. The hypothesis of this proposal is that strengthening problem solving skills among mothers of young children with ASDs serve as an important buffer against the negative impact of life stressors, and thereby prevent and attenuate depressive symptoms and parenting stress.

ELIGIBILITY:
Inclusion Criteria:

* all mothers of young children </ 6 with ASDs
* mothers who speak English or Spanish

Exclusion Criteria:

* Mother has psychosis
* Mother endorses suicidal ideation
* Mother actively using illicit drugs
* Mother expected to leave area within 6 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms | Baseline, 1.5, 3, 4.5, 6, 7.5 & 9 months
Parenting Stress Index | Baseline, 3, 6 & 9months
Perceived Stress Scale | Baseline, 3, 6 & 9 months

SECONDARY OUTCOMES:
Social Problem Solving Inventory | Baseline, 3, 6 & 9 months
Social Adjustment Scale Self-Report | Baseline, 3, 6 & 9 months
Patient Activation Measure | Baseline, 3, 6 & 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Feinberg E, Augustyn M, Fitzgerald E, Sandler J, Ferreira-Cesar Suarez Z, Chen N, Cabral H, Beardslee W, Silverstein M. Improving maternal mental health after a child's diagnosis of autism spectrum disorder: results from a randomized clinical trial. JAMA Pediatr. 2014 Jan;168(1):40-6. doi: 10.1001/jamapediatrics.2013.3445. PMID 24217336